CLINICAL TRIAL: NCT07107724
Title: Oxygen Consumption And Carbon Dioxide Production Following Hemodynamic Optimization In Shock: The OxyCarDio Study
Brief Title: O2 Consumption And CO2 Production After Hemodynamic Optimization In Shock
Acronym: OxyCarDio
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Antonio Maria Dell'Anna, Doctor, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7655
Record Dates: First submitted 2025-07-23; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamic Instability; Oxygen Consumption (V̇O2)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Noradrenalin — After inclusion, patients will be tested for fluid responsiveness. Pulse pressure variation (PPV) will be evaluated.
  In case of PPV> 13% a fluid bolus of 500 mL of Lactated Ringer's will be administered in 10 minutes.
  If PPV< 8% Norepinephrine will be administered or increased. If PPV is in the gray zone, a PLRT will be performed and if CO increases more than 10% a fluid bolus will be prescribed, otherwise norepinephrine increased.
Other: Fluid bolus — After inclusion, patients will be tested for fluid responsiveness. Pulse pressure variation (PPV) will be evaluated.
  In case of PPV> 13% a fluid bolus of 500 mL of Lactated Ringer's will be administered in 10 minutes.
  If PPV< 8% Norepinephrine will be administered or increased. If PPV is in the gray zone, a PLRT will be performed and if CO increases more than 10% a fluid bolus will be prescribed, otherwise norepinephrine increased.

SUMMARY:
The goal of this prospective observational study is to analyse change in VO2 and VCO2 measured via a dedicated ventilator after hemodynamic optimization maneuvers in adult patients admitted to the ICU with any sign of shock.

The main questions it aims to answer are:

1. Do common maneuvers for hemodynamic optimization (fluid bolus and/or vasopressor administration) have any impact on tissue perfusion in terms of oxygen consumption (VO2) and carbon dioxide production (VCO2) measured by a dedicated ventilator?
2. Are the values measured by exhaled gas comparable to those calculated by the measurement of dissolved veno-arterial gas?

Participants enrolled in the study will receive advanced hemodynamic monitoring with MostCare Up (Vygon ®) and their hemodynamic instability will be managed according to most recent guidelines and based on clinical decision of treating physicians.

ELIGIBILITY:
Inclusion Criteria:

Hypotension (MAP< 65mmHg or sudden drop in MAP > 15 mmHg) and one of the following conditions:

* Heart rate > 120 bpm
* Urinary output < 0.5 ml/kg/h for at least two hours
* Lactate > 2 mmol/L

Exclusion Criteria:

* Urgent need for surgery
* Urgent need for veno-arterial ECMO or severe hemodynamic instability
* Consistent risk of imminent death
* Severe ARDS or severe respiratory failure (p/F < 100 mmHg) and/or FiO2>0.8
* Severe heart failure (NYHA 4 and/or EF<25%)
* Need for intermittent or continuous renal replacement therapy (IRRT or CRRT)
* Anemia defined as Hb<8 g/dL
* VO2 variability < 5% throughout ten minutes of stabilization before procedure start
* Intraabdominal hypertension, defined as intraabdominal pressure > 18 mmHg
* Pregnancy
* Withdrawal or refuse of informed consent
* Terminal disease
* Do-not-resuscitate order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with signs of hemodynamic instability
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in VO2 | Two minutes after the end of fluid bolus infusion or vasopressor increase, and every 10 minutes for one hour
  Change in VO2, measured via a dedicated ventilator after either fluid expansion or increase in vasopressors administration.

SECONDARY OUTCOMES:
Change in VCO2 | Two minutes after the end of fluid bolus infusion or vasopressor increase, and every 10 minutes for one hour
  Change in VCO2, measured via a dedicated ventilator after either fluid expansion or increase in vasopressors administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario Fondazione Agostino Gemelli IRCCS, Roma, Italy